CLINICAL TRIAL: NCT04858789
Title: Effectiveness of a Culturally Adapted Cognitive Behavioral Intervention to Reducing Psychological Distress and Improving Well-Being Among University Students During the COVID-19 Pandemic
Brief Title: The Effectiveness of a CA-CBI on Psychological Distress of University Students During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020.465.IRB3.184
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Psychological Distress; Well-being
Keywords: Culturally adapted; Covid-19; Psychological distress; University students; Well-being; Online intervention
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally Adapted Cognitive Behavioral Intervention (CA-CBI) (Experimental): The experimental group will receive an 8-session CA-CBI in an online group format.
  Interventions: Behavioral: Culturally Adapted Cognitive Behavioral Intervention (CA-CBI)
- Control (No Intervention): The control (care as usual) group will receive the information about freely available psychological support options. After all the measurements are completed, the control group will be able to receive CA-CBI, too.

INTERVENTIONS:
Behavioral: Culturally Adapted Cognitive Behavioral Intervention (CA-CBI) — CA-CBI is an intervention based on Culturally Adapted Cognitive Behavioral Therapy (CA-CBT) which was developed by Devon Hinton. This transdiagnostic intervention has a structured manual which can be culturally adapted and it will be used to decrease psychological distress and increase well-being by targeting cognitive and behavioral changes.
  Arms: Culturally Adapted Cognitive Behavioral Intervention (CA-CBI)

SUMMARY:
The effectiveness study for Culturally Adapted Cognitive Behavioral Intervention will be conducted with university students to measure if this intervention if effective for decreasing the university students' psychological distress and increase their well-being during the COVID-19 pandemic. Potential participants will be given an informed consent and included in a screening procedure to decide their eligibility. 100 participants (50 in experimental and 50 in control group-randomly assigned) who pass the screening procedure will be invited to the effectiveness study. The experimental group will receive an 8-session intervention while the control group will receive information about the freely available psychological support options. The measurements will be conducted three times; one week before, one week after and five weeks after the intervention.

DETAILED DESCRIPTION:
Rapid increase in the COVID-19 cases and COVID-19 related deaths were followed by several precautions including the daily usage of masks, social distancing, temporary closure of work places, government departments, schools and universities. Due to these adversities and necessary precautions, people experience psychological distress and symptoms of depression and anxiety during the pandemic. Research shows that university students are at risk for developing psychological distress and common mental health disorder symptoms, and providing psychological interventions for university students may decrease the mental health problems of the students. However, considering the social distancing, these interventions must be delivered online. There are some studies indicate that online interventions may be effective as face-to-face interventions. Considering the mental health support need that the university students have during COVID-19, addressing this need may be beneficial for the mental health of university students in these uncertain times. There are various studies that showed the effectiveness of various form of interventions and one of them is Culturally Adapted Cognitive Behavioral (CA-CB) intervention developed by Hinton. CA-CB interventions were tested with adolescents and women in Turkey and found to decrease the psychological symptoms of these people. CA-CB interventions are based on the cognitive behavioral approach's principles but also include emotion regulation techniques, mindfulness and stretching exercises.

The investigators propose to conduct a randomized controlled trial in which they aim to apply a preventive culturally adapted cognitive behavioral intervention (CA-CBI) which is adapted to university students and COVID-19 related stressors. After the adaptation process is completed, the investigators will distribute an online survey to university students for the recruitment. The university students who would like to participate in the intervention study and are eligible to participate will be included. The investigators will randomly assign them into two arms (control and CA-CBI) and then deliver CA-CBI in a group format to the intervention arm. The investigators will examine whether the psychological distress levels and common mental health problems of the students in the intervention arm is decreased compared to the control arm. The investigators will examine the study outcomes of the both arms at three times: Pre-assessment (1 week before the intervention), post-assessment (1 week after the intervention) and follow-up assessment (1 month after the post-assessment). A process evaluation according to the WHO will be completed with 5 study completers, 5 drop-outs and 2 facilitators to evaluate the feasibility of delivering CA-CBI.

Although the CA-CBI was delivered in Turkey to different populations before, it was not tested with university students yet. In addition, there are scarce publications on the online delivered group interventions and to our knowledge, there is neither such research conducted during the pandemic nor research about the efficacy of online synchronous interventions in Turkey. The investigators will contribute to the literature by adapting CA-CBI to the university students who are affected from COVID-19. In addition, they will also add to the literature on online interventions by delivering CA-CBI online in a group format.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or above
* Being a university student
* Scoring 16 or above on Kessler Psychological Distress Scale (K10)
* Scoring 14 or belove on Patient Health Questionnaire-9 (PHQ-9)

Exclusion Criteria:

* Being older than 30 years
* Imminent suicidal risk
* Living outside of Turkey
* Having any type of psychiatric disorder
* Receiving any specialized psychological or psychiatric treatment at the time of application to the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Comparison of changes of the Kessler-10 Psychological Distress Scale (K10) over time | Change from baseline (One week before the intervention) to follow-up assessment (13 weeks after the pre-assessment)]
  Kessler-10 Psychological Distress Scale is a 10-item scale that aims to measure the psychological distress. Each item is scored from 1 (none of the time) to 5 (all of the time) providing a range between 10 and 50. Higher scores indicate more severe psychological distress.

SECONDARY OUTCOMES:
Comparison of changes of the Patient Health Questionnaire-9 (PHQ-9) over time | Change from baseline (One week before the intervention) to follow-up assessment (13 weeks after the pre-assessment)]
  Patient Health Questionnaire is a 9-item questionnaire that aims to measure the depressive symptoms. Each item is scored from 0 (not at all) to 3 (nearly every day) providing a range between 0 and 27. Higher scores indicate more severe depressive symptoms.
Comparison of changes of the General Anxiety Disorder-7 (GAD-7) over time | Change from baseline (One week before the intervention) to follow-up assessment (13 weeks after the pre-assessment)
  General Anxiety Disorder-7 is a 7-item questionnaire that aims to measure anxiety symptoms. Each item is scored from 0 (not at all) to 3 (nearly every day) providing a range between 0 and 21. Higher scores indicate higher levels of anxiety symptoms
Comparison of changes of the PTSD Checklist for The Diagnostic and Statistical Manual of Mental Disorders 5 (DSM 5) (PCL-5) over time | Change from baseline (One week before the intervention) to follow-up assessment (13 weeks after the pre-assessment)
  The PTSD Checklist for DSM-5 is a 20-item questionnaire that assesses the symptoms of post-traumatic stress disorder. Each item is scored from 0 (not at all) to 4 (extremely) providing a range between 0 and 80. Higher scores indicate higher levels of PTSD symptoms.
Comparison of changes of the World Health Organization (Five) Well-Being Index (WHO-5) over time | Change from baseline (One week before the intervention) to follow-up assessment (13 weeks after the pre-assessment)
  The World Health Organization (Five) Well-Being Index (WHO-5) is a 5-item questionnaire that aims to measure well-being. Each item is scored from 0 (at no time) to 5 (all of the time) providing a range between 0 and 25. Higher scores indicate better well-being.

OTHER OUTCOMES:
Comparison of changes of the Dispositional Hope Scale over time | Change from baseline (One week before the intervention) to follow-up assessment (13 weeks after the pre-assessment)]
  The Dispositional Hope Scale is a 12-item questionnaire that aims to measure the dispositional hope. Each item is scored from 1 (definitely false) to 8 (definitely true) providing a range between 8 and 96. Higher scores indicate higher levels of dispositional hope.
Comparison of changes of the Emotion Regulation Questionnaire over time | Change from baseline (One week before the intervention) to follow-up assessment (13 weeks after the pre-assessment)]
  The Emotion Regulation Questionnaire is a 10-item questionnaire that aims to measure individual differences in emotion regulation and its strategies. Each item is scored from 1 (strongly disagree) to 7 (strongly agree) providing a range between 10 and 70. It has two subscales which are re-appraisal and suppression. Higher scores indicate more frequent use of these strategies.
8. Comparison of changes of the Acceptance and Action Questionnaire-II (AAQ-II) over time | Change from baseline (One week before the intervention) to follow-up assessment (13 weeks after the pre-assessment)
  The Acceptance and Action Questionnaire-II is a 7-item questionnaire that aims to measure psychological flexibility. Each item is scored from 1 (never true) to 7 (always true) providing a range between 7 and 49. Higher scores indicate less psychological flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Ekin Çakır, PhD Student, Study Chair — Koç University
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hinton DE, Chhean D, Pich V, Safren SA, Hofmann SG, Pollack MH. A randomized controlled trial of cognitive-behavior therapy for Cambodian refugees with treatment-resistant PTSD and panic attacks: a cross-over design. J Trauma Stress. 2005 Dec;18(6):617-29. doi: 10.1002/jts.20070. PMID 16382423
- [Background] Hinton DE, Pham T, Tran M, Safren SA, Otto MW, Pollack MH. CBT for Vietnamese refugees with treatment-resistant PTSD and panic attacks: a pilot study. J Trauma Stress. 2004 Oct;17(5):429-33. doi: 10.1023/B:JOTS.0000048956.03529.fa. PMID 15633922
- [Background] Huang J, Nigatu YT, Smail-Crevier R, Zhang X, Wang J. Interventions for common mental health problems among university and college students: A systematic review and meta-analysis of randomized controlled trials. J Psychiatr Res. 2018 Dec;107:1-10. doi: 10.1016/j.jpsychires.2018.09.018. Epub 2018 Sep 29. PMID 30300732
- [Background] Vindegaard N, Benros ME. COVID-19 pandemic and mental health consequences: Systematic review of the current evidence. Brain Behav Immun. 2020 Oct;89:531-542. doi: 10.1016/j.bbi.2020.05.048. Epub 2020 May 30. PMID 32485289
- [Background] Carlbring P, Andersson G, Cuijpers P, Riper H, Hedman-Lagerlof E. Internet-based vs. face-to-face cognitive behavior therapy for psychiatric and somatic disorders: an updated systematic review and meta-analysis. Cogn Behav Ther. 2018 Jan;47(1):1-18. doi: 10.1080/16506073.2017.1401115. Epub 2017 Dec 7. PMID 29215315
- [Background] Cao W, Fang Z, Hou G, Han M, Xu X, Dong J, Zheng J. The psychological impact of the COVID-19 epidemic on college students in China. Psychiatry Res. 2020 May;287:112934. doi: 10.1016/j.psychres.2020.112934. Epub 2020 Mar 20. PMID 32229390
- [Background] Acarturk ZC, Abuhamdeh S, Jalal B, Unaldi N, Alyanak B, Cetinkaya M, Gulen B, Hinton D. Culturally adapted transdiagnostic CBT for SSRI resistant Turkish adolescents: A pilot study. Am J Orthopsychiatry. 2019;89(2):222-227. doi: 10.1037/ort0000310. Epub 2018 Jan 18. PMID 29345479

DOCUMENTS (2):
  • Study Protocol (2021-03-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT04858789/Prot_000.pdf
  • Informed Consent Form (2021-03-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT04858789/ICF_001.pdf